CLINICAL TRIAL: NCT00838903
Title: A Randomized, Double-Blind, Placebo and Active-Controlled, Parallel-Group, Multicenter Study to Determine the Efficacy and Safety of Albiglutide When Used in Combination With Metformin Compared With Metformin Plus Sitagliptin, Metformin Plus Glimepiride, and Metformin Plus Placebo in Subjects With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Albiglutide in Treatment of Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112753
Record Dates: First submitted 2009-02-05; First posted 2009-02-09 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — rGLP-1 protein; Sitagliptin Phosphate; glimepiride; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- albiglutide + metformin (Experimental): Albiglutide + metformin + placebo sitagliptin + placebo glimepiride
  Interventions: Biological: albiglutide; Drug: metformin; Drug: placebo sitagliptin; Drug: placebo glimepiride
- sitagliptin + metformin (Active Comparator): Sitagliptin + metformin + placebo albiglutide + placebo glimepiride
  Interventions: Drug: sitagliptin; Drug: metformin; Biological: placebo albiglutide; Drug: placebo glimepiride
- glimepiride + metformin (Active Comparator): Glimepiride + metformin + placebo albiglutide + placebo sitagliptin
  Interventions: Drug: glimepiride; Drug: metformin; Biological: placebo albiglutide; Drug: placebo sitagliptin
- metformin + placebo (Active Comparator): Metformin + placebo albiglutide + placebo sitagliptin + placebo glimepiride
  Interventions: Drug: metformin; Biological: placebo albiglutide; Drug: placebo sitagliptin; Drug: placebo glimepiride

INTERVENTIONS:
Biological: albiglutide — albiglutide
  Arms: albiglutide + metformin
Drug: sitagliptin — sitagliptin
  Arms: sitagliptin + metformin
Drug: glimepiride — Glimepiride
  Arms: glimepiride + metformin
Drug: metformin — Metformin
Biological: placebo albiglutide — placebo to match albiglutide
  Arms: glimepiride + metformin; metformin + placebo; sitagliptin + metformin
Drug: placebo sitagliptin — placebo to match sitagliptin
  Arms: albiglutide + metformin; glimepiride + metformin; metformin + placebo
Drug: placebo glimepiride — placebo to match glimepiride
  Arms: albiglutide + metformin; metformin + placebo; sitagliptin + metformin

SUMMARY:
The purpose of this study is to determine if albiglutide is safe and effective in the treatment of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* BMI 20-45kg/m2 inclusive

Exclusion Criteria:

* females who are pregnant, lactating or <6 weeks post-partum
* current symptomatic heart failure (NYHA Class III or IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1049 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (322):
- United States (257):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Hueytown, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Green Valley, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Bull Shoals, Arkansas
  - GSK Investigational Site, Harrisburg, Arkansas
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Searcy, Arkansas
  - GSK Investigational Site, Buena Park, California
  - GSK Investigational Site, Carmichael, California
  - GSK Investigational Site, Chino, California
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Escondido, California
  - GSK Investigational Site, Foothill Ranch, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Indio, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Lakewood, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Alamitos, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Palm Desert, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Satna Monica, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Victorville, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Arvada, Colorado
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Trumbull, Connecticut
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Middletown, Delaware
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Cutler Bay, Florida
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Lauderdale Lakes, Florida
  - GSK Investigational Site, Marianna, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Oviedo, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Ponte Vedra Beach, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Snellville, Georgia
  - GSK Investigational Site, Stone Mountain, Georgia
  - GSK Investigational Site, Tucker, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Aurora, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evergreen Park, Illinois
  - GSK Investigational Site, La Grange, Illinois
  - GSK Investigational Site, Naperville, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Fishers, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, La Porte, Indiana
  - GSK Investigational Site, Muncie, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Dubuque, Iowa
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Waterloo, Iowa
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Mission, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Crescent Springs, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Hyattsville, Maryland
  - GSK Investigational Site, Oxon Hill, Maryland
  - GSK Investigational Site, Haverhill, Massachusetts
  - GSK Investigational Site, Bay City, Michigan
  - GSK Investigational Site, Benzonia, Michigan
  - GSK Investigational Site, Cadillac, Michigan
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Interlochen, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Saint Clair Shores, Michigan
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, Picayune, Mississippi
  - GSK Investigational Site, Rolling Fork, Mississippi
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, West Plains, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Great Falls, Montana
  - GSK Investigational Site, Broken Bow, Nebraska
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Berlin, New Jersey
  - GSK Investigational Site, Elizabeth, New Jersey
  - GSK Investigational Site, Haddon Heights, New Jersey
  - GSK Investigational Site, Hainesport, New Jersey
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Stratford, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, North Massapequa, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Asheboro, North Carolina
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Burlington, North Carolina
  - GSK Investigational Site, Calabash, North Carolina
  - GSK Investigational Site, Chadbourn, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Lenoir, North Carolina
  - GSK Investigational Site, Mint Hill, North Carolina
  - GSK Investigational Site, Morehead City, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Tabor City, North Carolina
  - GSK Investigational Site, Grand Forks, North Dakota
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Canal Fulton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Mason, Ohio
  - GSK Investigational Site, Maumee, Ohio
  - GSK Investigational Site, Thornville, Ohio
  - GSK Investigational Site, Zanesville, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Ashland, Oregon
  - GSK Investigational Site, Bensalem, Pennsylvania
  - GSK Investigational Site, Carlisle, Pennsylvania
  - GSK Investigational Site, Downington, Pennsylvania
  - GSK Investigational Site, Feasterville, Pennsylvania
  - GSK Investigational Site, Harrisburg, Pennsylvania
  - GSK Investigational Site, Landsdale, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Tipton, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Cumberland, Rhode Island
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Manning, South Carolina
  - GSK Investigational Site, Murrells Inlet, South Carolina
  - GSK Investigational Site, North Myrtle Beach, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Taylors, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Columbia, Tennessee
  - GSK Investigational Site, Fayetteville, Tennessee
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, McKenzie, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Tullahoma, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Cleburne, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Deer Park, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Hurst, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Lake Jackson, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, North Richland Hills, Texas
  - GSK Investigational Site, Odessa, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Schertz, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Sugarland, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, West Valley City, Utah
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Suffolk, Virginia
  - GSK Investigational Site, Virgina Beach, Virginia
  - GSK Investigational Site, Weber City, Virginia
  - GSK Investigational Site, Federal Way, Washington
  - GSK Investigational Site, Richland, Washington
  - GSK Investigational Site, Selah, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Lewisburg, West Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin
- GSK Investigational Site, Alabaster, Albania
- Germany (7):
  - GSK Investigational Site, Villingen-Schwenningen, Baden-Wurttemberg
  - GSK Investigational Site, Kelkheim, Hesse
  - GSK Investigational Site, Rotenburg an der Fulda, Hesse
  - GSK Investigational Site, Bad Lauterberg im Harz, Lower Saxony
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Berlin, State of Berlin
- Hong Kong (3):
  - GSK Investigational Site, Kwun Tong, Kowloon
  - GSK Investigational Site, Shatin
  - GSK Investigational Site, Tai Po
- Mexico (14):
  - GSK Investigational Site, Tijuana, Baja California Norte
  - GSK Investigational Site, Torreón, Coahuila
  - GSK Investigational Site, Durango, Durango
  - GSK Investigational Site, Pachuca, Hidalgo
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Morelia, Michoacán
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Puebla City, Puebla
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Distrito Federal
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Nezahualcóyotl
- Peru (4):
  - GSK Investigational Site, Ica, Ica
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Callao, Lima
  - GSK Investigational Site, Piura, Piura
- Philippines (4):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, San Juan City
  - GSK Investigational Site, Taytay Rizal
- Russia (7):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Yaroslavl
- South Africa (12):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Boksburg North, Gauteng
  - GSK Investigational Site, Johannesburg, Gauteng
  - GSK Investigational Site, Lenasia, Gauteng
  - GSK Investigational Site, Parktown, Gauteng
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Kempton Park
  - GSK Investigational Site, Parow
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Soweto
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Seville
- United Kingdom (11):
  - GSK Investigational Site, Plymouth, Devon
  - GSK Investigational Site, Canterbury, Kent
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Sunbury-on-Thames, Middlesex
  - GSK Investigational Site, Port Glasgow, Renfrewshire
  - GSK Investigational Site, Coventry, West Midlands
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Hull
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Home PD, Ahren B, Reusch JEB, Rendell M, Weissman PN, Cirkel DT, Miller D, Ambery P, Carr MC, Nauck MA. Three-year data from 5 HARMONY phase 3 clinical trials of albiglutide in type 2 diabetes mellitus: Long-term efficacy with or without rescue therapy. Diabetes Res Clin Pract. 2017 Sep;131:49-60. doi: 10.1016/j.diabres.2017.06.013. Epub 2017 Jun 15. PMID 28683300
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 112753 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112753 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112753 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112753 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112753 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112753 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112753 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants (par.) entered a 2-week Screening Period, a 4-week Run-in/Stabilization Period, a 156-week Treatment Period, and a 8-week post-treatment Follow-up Period. A total of 1525 par. were screened, 1049 were randomized and 1012 par. received at least 1 dose of study treatment.
Groups:
- Placebo Plus Metformin: Participants received metformin >=1500 milligrams (mg) daily plus matching albiglutide placebo as a subcutaneous injection weekly via a fully disposable pen injector system plus matching sitagliptin placebo plus matching glimepiride placebo from Week 1 to Week 156. All participants returned for the 8-week post-treatment Follow-up Period.
- Sitagliptin 100 mg Plus Metformin: Participants received sitagliptin 100 mg daily plus metformin >=1500 mg daily plus matching albiglutide placebo as a subcutaneous injection weekly via a fully disposable pen injector system plus matching glimepiride placebo from Week 1 to Week 156. All participants returned for the 8-week post-treatment Follow-up Period.
- Glimepiride 2 mg Plus Metformin: Participants received glimepiride 2 mg daily (with masked up-titration to 4 mg daily if required) plus metformin >=1500 mg daily plus matching albiglutide placebo as a subcutaneous injection weekly via a fully disposable pen injector system plus matching sitagliptin placebo from Week 1 to Week 156. All participants returned for the 8-week post-treatment Follow-up Period.
- Albiglutide 30 mg Plus Metformin: Participants received albiglutide 30 mg weekly (with masked up-titration to 50 mg weekly if required) as a subcutaneous injection via a fully disposable pen injector system plus metformin >=1500 mg daily plus matching sitagliptin placebo plus matching glimepiride placebo from Week 1 to Week 156. All participants returned for the 8-week post-treatment Follow-up Period.
Period: Treatment Period (156 Weeks)
Arm/Group | Placebo Plus Metformin | Sitagliptin 100 mg Plus Metformin | Glimepiride 2 mg Plus Metformin | Albiglutide 30 mg Plus Metformin
Started | 101 | 302 | 307 | 302
Missing Active Treatment Status | 1 | 0 | 0 | 0
Completed | 55 | 190 | 191 | 192
Not Completed | 46 | 112 | 116 | 110
Not completed — Adverse Event | 5 | 13 | 17 | 25
Not completed — Protocol Violation | 1 | 6 | 6 | 5
Not completed — Noncompliance | 9 | 13 | 12 | 6
Not completed — Severe or Repeated Hypoglycaemia | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 4 | 16 | 15 | 13
Not completed — Withdrawal by Subject | 20 | 55 | 56 | 53
Not completed — Physician Decision | 1 | 2 | 1 | 2
Not completed — Termination of Study/Site by GSK | 3 | 5 | 5 | 4
Not completed — Patient and PI Decision to Discontinue | 0 | 1 | 0 | 0
Not completed — Poor Glycemic Control | 0 | 0 | 0 | 1
Not completed — Poor Therapeutic Response | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — PI Decided for Safety Purpose | 0 | 0 | 1 | 0
Not completed — Site closed | 0 | 0 | 1 | 0
Not completed — Site Closed and Subject Withdrew Consent | 1 | 0 | 0 | 0
Not completed — Subject Migrated to Other Country | 0 | 1 | 0 | 1
Not completed — Missing Active Treatment Status | 1 | 0 | 0 | 0
Period: Follow-up Period (8 Weeks)
Arm/Group | Placebo Plus Metformin | Sitagliptin 100 mg Plus Metformin | Glimepiride 2 mg Plus Metformin | Albiglutide 30 mg Plus Metformin
Started | 101 (Participants withdrawing from the Treatment Period entered the Follow-up Period.) | 302 (Participants withdrawing from the Treatment Period entered the Follow-up Period.) | 307 (Participants withdrawing from the Treatment Period entered the Follow-up Period.) | 302 (Participants withdrawing from the Treatment Period entered the Follow-up Period.)
Completed | 75 | 237 | 243 | 244
Not Completed | 26 | 65 | 64 | 58
Not completed — Adverse Event | 0 | 0 | 3 | 1
Not completed — Noncompliance | 2 | 8 | 5 | 5
Not completed — Lost to Follow-up | 6 | 28 | 22 | 24
Not completed — Did Not Enter Follow-up Period | 5 | 7 | 12 | 7
Not completed — Subject Withdrawn from Follow-up | 8 | 13 | 14 | 14
Not completed — Physician Decision | 1 | 1 | 1 | 1
Not completed — Termination of Study/Site by GSK | 3 | 4 | 6 | 4
Not completed — ICF Withdrawn | 0 | 1 | 0 | 0
Not completed — Investigator Stopped Study at Site | 0 | 1 | 0 | 0
Not completed — Subject Moved out of Town | 0 | 0 | 0 | 1
Not completed — Missing | 1 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Metformin | Sitagliptin 100 mg Plus Metformin | Glimepiride 2 mg Plus Metformin | Albiglutide 30 mg Plus Metformin | Total
Number analyzed (Participants) | 101 | 302 | 307 | 302 | 1012
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.1 (10.01) | 54.3 (9.81) | 54.4 (9.97) | 54.3 (10.12) | 54.5 (9.97)
Gender [Count of Participants; unit: Participants]
  Female | 51 | 163 | 149 | 167 | 530
  Male | 50 | 139 | 158 | 135 | 482
Race/Ethnicity, Customized [Number; unit: Participants] — A participant may have been counted in more than one category.
  Participants
    African American/African Heritage | 23 | 35 | 39 | 53 | 150
    American Indian or Alaskan Native | 9 | 22 | 25 | 17 | 73
    Asian - Central/South Asian Heritage | 1 | 7 | 3 | 2 | 13
    Asian - East Asian Heritage | 0 | 2 | 3 | 5 | 10
    Asian - Japanese Heritage | 1 | 0 | 1 | 0 | 2
    Asian - South East Asian Heritage | 3 | 11 | 9 | 11 | 34
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 2
    White - Arabic/North African Heritage | 0 | 1 | 9 | 3 | 13
    White - White/Caucasian/European Heritage | 64 | 225 | 220 | 214 | 723

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Glycosylated Hemoglobin (HbA1c) at Week 104
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The BL HbA1c value is defined as the last non-missing value before the start of treatment. Change from BL was calculated as the value at Week 104 minus the value at BL. Based on analysis of covariance (ANCOVA): change = treatment + BL HbA1c + prior myocardial infarction history + age category + region. Difference of least squares means (albiglutide - placebo, albiglutide - sitagliptin, albiglutide - glimepiride) is from the ANCOVA model. The last observation carried forward (LOCF) method was used to impute missing post-Baseline HbA1c values; the last non-missing post-BL on-treatment measurement was used to impute the missing measurement. HbA1c values obtained after hyperglycemic rescue were treated as missing and were replaced with pre-rescue values.
Time Frame: Baseline and Week 104
Population: Intent-to-Treat (ITT) Population with LOCF: all randomized par. who received >=1 dose of study medication and who had a BL assessment and >=1 post-BL assessment of HbA1c. Only par. with a value at BL and at the specified visit were analyzed. Values were carried forward for par. who were rescued or discontinued from active treatment before Week 104.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c in the blood
Arm/Group | Placebo Plus Metformin | Sitagliptin 100 mg Plus Metformin | Glimepiride 2 mg Plus Metformin | Albiglutide 30 mg Plus Metformin
Number analyzed (Participants) | 97 | 297 | 299 | 293
Percentage of HbA1c in the blood | 0.27 (0.113) | -0.28 (0.065) | -0.36 (0.064) | -0.63 (0.065)
Statistical Analysis 1: Comparison: Placebo Plus Metformin vs Albiglutide 30 mg Plus Metformin; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -0.91, 95% CI 2-sided [-1.16 to -0.65]
Statistical Analysis 2: Comparison: Sitagliptin 100 mg Plus Metformin vs Albiglutide 30 mg Plus Metformin; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -0.35, 95% CI 2-sided [-0.53 to -0.17]
Statistical Analysis 3: Comparison: Glimepiride 2 mg Plus Metformin vs Albiglutide 30 mg Plus Metformin; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.45 to -0.09]
Statistical Analysis 4: Comparison: Placebo Plus Metformin vs Albiglutide 30 mg Plus Metformin; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — The p-value is for superiority testing of albiglutide over placebo at 0.05 level; The p-value is from a two-sided t-test to test whether the difference of least square means (albiglutide - placebo) is equal to zero
Statistical Analysis 5: Comparison: Sitagliptin 100 mg Plus Metformin vs Albiglutide 30 mg Plus Metformin; Test type: Non-Inferiority or Equivalence — To test whether the difference of least square means (albiglutide - sitagliptin) is equal to the pre-specified non-inferiority margin of 0.3%; p < 0.0001, t-test, 1 sided — The p-value is for non-inferiority testing of albiglutide versus sitagliptin at 0.0125 level
Statistical Analysis 6: Comparison: Glimepiride 2 mg Plus Metformin vs Albiglutide 30 mg Plus Metformin; Test type: Non-Inferiority or Equivalence — To test whether the difference of least square means (albiglutide - glimepiride) is equal to the pre-specified non-inferiority margin of 0.3%; p < 0.0001, t-test, 1 sided — The p-value is for non-inferiority testing of albiglutide versus glimepiride at 0.0125 level
Statistical Analysis 7: Comparison: Sitagliptin 100 mg Plus Metformin vs Albiglutide 30 mg Plus Metformin; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided — The p-value is for superiority testing of albiglutide versus sitagliptin at 0.025 level; The p-value is from a two-sided t-test to test whether the difference of least square means (albiglutide - sitagliptin) is equal to zero
Statistical Analysis 8: Comparison: Glimepiride 2 mg Plus Metformin vs Albiglutide 30 mg Plus Metformin; Test type: Superiority or Other; p = 0.0033, t-test, 2 sided — The p-value is for superiority testing of albiglutide versus glimepiride at 0.025 level; The p-value is from a two-sided t-test to test whether the difference of least square means (albiglutide - glimepiride) is equal to zero

2. Secondary Outcome: Change From Baseline in HbA1c at Week 156
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. This analysis used observed HbA1c values, excluding those obtained after hyperglycemia rescue; no missing data imputation was performed .
Time Frame: Baseline and Week 156
Population: Intent-to-Treat (ITT) Population with observed values. Only those par. with a value at Baseline and at the specified visit were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in the blood
Arm/Group | Placebo Plus Metformin | Sitagliptin 100 mg Plus Metformin | Glimepiride 2 mg Plus Metformin | Albiglutide 30 mg Plus Metformin
Number analyzed (Participants) | 16 | 88 | 102 | 115
Percentage of HbA1c in the blood | -0.46 (0.820) | -0.56 (1.160) | -0.59 (0.999) | -0.88 (0.959)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 104
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is the last non-missing value before the start of treatment. The LOCF method was used to impute missing post-Baseline FPG values. FPG values obtained after hyperglycemia rescue were treated as missing and replaced with pre-rescue values. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Based on ANCOVA: change = treatment + Baseline FPG + Baseline HbA1c category + prior myocardial infarction history + age category + region.
Time Frame: Baseline and Week 104
Population: Intent-to-Treat (ITT) Population with LOCF. Only those participants with a value at Baseline and at the specified visit were analyzed. Values were carried forward for participants who were rescued or discontinued from active treatment before Week 104.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo Plus Metformin | Sitagliptin 100 mg Plus Metformin | Glimepiride 2 mg Plus Metformin | Albiglutide 30 mg Plus Metformin
Number analyzed (Participants) | 100 | 299 | 302 | 296
Millimoles per liter (mmol/L) | 0.55 (0.277) | -0.12 (0.160) | -0.41 (0.159) | -0.98 (0.161)

4. Secondary Outcome: Change From Baseline in FPG at Week 156
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. This analysis used observed FPG values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline and Week 156
Population: ITT Population with observed values. Only those participants with a value at Baseline and at the specified visit were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo Plus Metformin | Sitagliptin 100 mg Plus Metformin | Glimepiride 2 mg Plus Metformin | Albiglutide 30 mg Plus Metformin
Number analyzed (Participants) | 16 | 88 | 98 | 112
Millimoles per liter (mmol/L) | -0.11 (1.498) | -0.50 (2.519) | -0.71 (2.684) | -1.30 (2.602)

5. Secondary Outcome: Number of Participants Who Achieved Clinically Meaningful HbA1c Response Levels of <6.5%, <7%, and <7.5% at Week 104
Description: The number of participants who achieved the HbA1c treatment goal (i.e., HbA1c response levels of <6.5%, <7%, and <7.5% at Week 52) were assessed.
Time Frame: Week 104
Population: ITT Population with LOCF. Only those participants with a value at Baseline and at the specified visit were analyzed. Values were carried forward for participants who were rescued or discontinued from active treatment before Week 104.
Measure: Number; unit: Participants
Arm/Group | Placebo Plus Metformin | Sitagliptin 100 mg Plus Metformin | Glimepiride 2 mg Plus Metformin | Albiglutide 30 mg Plus Metformin
Number analyzed (Participants) | 97 | 297 | 299 | 293
Participants
  HbA1c <6.5% | 7 | 45 | 40 | 50
  HbA1c <7.0% | 15 | 94 | 94 | 113
  HbA1c <7.5% | 27 | 132 | 147 | 172

6. Secondary Outcome: Number of Participants Who Achieved Clinically Meaningful HbA1c Response Levels of <6.5%, <7%, and <7.5% at Week 156
Description: The number of participants who achieved the HbA1c treatment goal (i.e., HbA1c response levels of <6.5%, <7%, and <7.5% at Week 156) were assessed.
Time Frame: Week 156
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Placebo Plus Metformin | Sitagliptin 100 mg Plus Metformin | Glimepiride 2 mg Plus Metformin | Albiglutide 30 mg Plus Metformin
Number analyzed (Participants) | 16 | 88 | 102 | 115
Participants
  HbA1c <6.5% | 4 | 23 | 15 | 31
  HbA1c <7.0% | 7 | 44 | 44 | 69
  HbA1c <7.5% | 13 | 69 | 69 | 90

7. Secondary Outcome: Time to Hyperglycemia Rescue
Description: Participants who experienced persistent hyperglycemia (high blood glucose) could have qualified for hyperglycemia rescue.The conditions for hyperglycemic rescue were as follows: FPG >=280 milligrams/deciliter (mg/dL) between >=Week 2 and <Week 4; FPG >=250 mg/dL between >=Week 4 and <Week 12; HbA1c >=8.5% and a <=0.5% reduction from Baseline between >=Week 12 and <Week 24; HbA1c >=8.5% between >=Week 24 and <Week 48; HbA1c >=8.0% between >= Week 48 and <Week 156. Participants could have been rescued at any time on or after Week 2. Time to hyperglycemia rescue is defined as the time between the date of the first dose of study medication and the date of hyperglycemia rescue plus 1 day, or the time between the date of the first dose of study medication and the date of the last visit during the active treatment period plus 1 day for participants not requiring rescue. This time was divided by 7 to express the result in week
Time Frame: From the start of study medication until the end of the treatment (up to Week 156)
Population: ITT Population. Only those participants with a value at Baseline and at the specified visit were analyzed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo Plus Metformin | Sitagliptin 100 mg Plus Metformin | Glimepiride 2 mg Plus Metformin | Albiglutide 30 mg Plus Metformin
Number analyzed (Participants) | 100 | 300 | 302 | 297
Weeks | 67.71 [53.14 to 122.14] | NA [NA to NA] — There were few events of hyperglycemia rescue (<50% of participants with events) to calculate the median and confidence interval. | NA [NA to NA] — There were few events of hyperglycemia rescue (<50% of participants with events) to calculate the median and confidence interval. | NA [NA to NA] — There were few events of hyperglycemia rescue (<50% of participants with events) to calculate the median and confidence interval.

8. Secondary Outcome: Change From Baseline in Body Weight at Week 104
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight. The LOCF method was used to impute missing post-Baseline weight values. Weight values obtained after hyperglycemia rescue were treated as missing and replaced with prerescue values. Based on ANCOVA: change = treatment + Baseline weight + Baseline HbA1c category + prior myocardial infarction history + age category + region.
Time Frame: Baseline and Week 104
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo Plus Metformin | Sitagliptin 100 mg Plus Metformin | Glimepiride 2 mg Plus Metformin | Albiglutide 30 mg Plus Metformin
Number analyzed (Participants) | 100 | 300 | 302 | 296
Kilograms | -1.00 (0.411) | -0.86 (0.237) | 1.17 (0.237) | -1.21 (0.239)

9. Secondary Outcome: Change From Baseline in Body Weight at Week 156
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight. This analysis used observed body weight values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline and Week 156
Population: ITT Population with observed values. Only those participants who were available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Placebo Plus Metformin | Sitagliptin 100 mg Plus Metformin | Glimepiride 2 mg Plus Metformin | Albiglutide 30 mg Plus Metformin
Number analyzed (Participants) | 16 | 89 | 102 | 116
Kilograms | -3.61 (3.460) | -2.05 (4.109) | 0.98 (4.760) | -2.31 (5.093)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs, defined as those events that had a start date on or after the first day of study medication and within 56 days after the end of study medication (up to Week 156), are reported.
Description: SAEs and non-serious AEs are reported for members of the Safety Population, comprised of all participants who received at least one dose of study treatment.
Arm/Group | Placebo Plus Metformin | Sitagliptin 100 mg Plus Metformin | Glimepiride 2 mg Plus Metformin | Albiglutide 30 mg Plus Metformin
Serious Adverse Events (participants affected / at risk) | 15/101 | 32/302 | 36/307 | 44/302
Other Adverse Events (participants affected / at risk) | 75/101 | 229/302 | 258/307 | 242/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Metformin (N=101) | Sitagliptin 100 mg Plus Metformin (N=302) | Glimepiride 2 mg Plus Metformin (N=307) | Albiglutide 30 mg Plus Metformin (N=302)
Pneumonia (Infections and infestations) | 1 | 2 | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 3
Pyelonephritis acute (Infections and infestations) | 1 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 2 | 1 | 2
Coronary artery disease (Cardiac disorders) | 2 | 1 | 2 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 2
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 2 | 4
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 1
Device malfunction (General disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0
Complicated migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Viith nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
Ischaemia (Vascular disorders) | 0 | 1 | 0 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 1 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Cervical Polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Metformin (N=101) | Sitagliptin 100 mg Plus Metformin (N=302) | Glimepiride 2 mg Plus Metformin (N=307) | Albiglutide 30 mg Plus Metformin (N=302)
Upper respiratory tract infection (Infections and infestations) | 10 | 33 | 32 | 58
Urinary tract infection (Infections and infestations) | 11 | 37 | 35 | 27
Nasopharyngitis (Infections and infestations) | 9 | 31 | 30 | 24
Bronchitis (Infections and infestations) | 10 | 26 | 23 | 24
Influenza (Infections and infestations) | 7 | 17 | 25 | 21
Gastroenteritis (Infections and infestations) | 4 | 16 | 9 | 19
Pharyngitis (Infections and infestations) | 10 | 22 | 17 | 17
Sinusitis (Infections and infestations) | 5 | 22 | 22 | 17
Herpes zoster (Infections and infestations) | 1 | 2 | 5 | 8
Cellulitis (Infections and infestations) | 1 | 7 | 6 | 7
Pneumonia (Infections and infestations) | 1 | 2 | 7 | 6
Tooth abscess (Infections and infestations) | 6 | 10 | 7 | 4
Otitis media (Infections and infestations) | 1 | 7 | 2 | 4
Ear infection (Infections and infestations) | 3 | 5 | 6 | 3
Viral infection (Infections and infestations) | 1 | 7 | 4 | 3
Lower respiratory tract infection (Infections and infestations) | 4 | 6 | 1 | 3
Gastroenteritis viral (Infections and infestations) | 1 | 7 | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 28 | 31 | 46
Nausea (Gastrointestinal disorders) | 13 | 22 | 25 | 37
Vomiting (Gastrointestinal disorders) | 1 | 14 | 13 | 22
Constipation (Gastrointestinal disorders) | 14 | 8 | 13 | 19
Dyspepsia (Gastrointestinal disorders) | 2 | 5 | 8 | 13
Abdominal pain (Gastrointestinal disorders) | 0 | 12 | 8 | 12
Gastritis (Gastrointestinal disorders) | 4 | 7 | 7 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 10 | 10 | 7
Abdominal pain upper (Gastrointestinal disorders) | 3 | 6 | 3 | 4
Flatulence (Gastrointestinal disorders) | 3 | 1 | 1 | 4
Dental caries (Gastrointestinal disorders) | 3 | 7 | 8 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 7 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 31 | 28 | 24
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 11 | 6 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 22 | 19 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 15 | 21 | 17
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 11 | 9 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 8 | 9 | 10
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 5 | 3 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 5 | 6
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 7 | 4
Hypoglycaemia (Musculoskeletal and connective tissue disorders) | 18 | 24 | 102 | 35
Dyslipidaemia (Metabolism and nutrition disorders) | 4 | 11 | 5 | 9
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 8 | 12 | 8
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 4 | 6 | 7
Gout (Metabolism and nutrition disorders) | 2 | 3 | 3 | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 4 | 7 | 3
Headache (Nervous system disorders) | 5 | 26 | 34 | 22
Dizziness (Nervous system disorders) | 5 | 13 | 14 | 10
Neuropathy peripheral (Nervous system disorders) | 1 | 5 | 7 | 8
Diabetic neuropathy (Nervous system disorders) | 2 | 5 | 7 | 5
Paraesthesia (Nervous system disorders) | 3 | 3 | 5 | 4
Sciatica (Nervous system disorders) | 3 | 1 | 1 | 2
Amnesia (Nervous system disorders) | 3 | 0 | 1 | 1
Injection site reaction (General disorders) | 2 | 5 | 9 | 33
Oedema peripheral (General disorders) | 2 | 10 | 25 | 13
Injection site haematoma (General disorders) | 2 | 11 | 11 | 9
Fatigue (General disorders) | 4 | 8 | 6 | 8
Chest pain (General disorders) | 3 | 6 | 5 | 8
Injection site erythema (General disorders) | 1 | 2 | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 24 | 28 | 26
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 16 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 10 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 9 | 4
Hypertension (Vascular disorders) | 6 | 28 | 32 | 32
Diabetic retinopathy (Eye disorders) | 2 | 7 | 14 | 14
Cataract (Eye disorders) | 6 | 12 | 20 | 13
Conjunctivitis (Eye disorders) | 0 | 4 | 7 | 4
Depression (Psychiatric disorders) | 5 | 9 | 10 | 15
Insomnia (Psychiatric disorders) | 2 | 6 | 10 | 12
Anxiety (Psychiatric disorders) | 6 | 6 | 9 | 8
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 7 | 8
Excoriation (Injury, poisoning and procedural complications) | 2 | 2 | 5 | 7
Muscle strain (Injury, poisoning and procedural complications) | 4 | 4 | 9 | 6
Fall (Injury, poisoning and procedural complications) | 1 | 7 | 0 | 6
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 8 | 9 | 5
Anaemia (Blood and lymphatic system disorders) | 8 | 14 | 12 | 14
Rash (Skin and subcutaneous tissue disorders) | 0 | 8 | 5 | 10
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 0
Seasonal allergy (Immune system disorders) | 1 | 3 | 5 | 8
Erectile Dysfunction (Reproductive system and breast disorders) | 3 | 4 | 4 | 6
Vertigo (Ear and labyrinth disorders) | 3 | 3 | 1 | 8
Weight Increased (Investigations) | 1 | 2 | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.